CLINICAL TRIAL: NCT05889169
Title: Stroke-induced Immunodepression: Role in the Neurorehabilitation Setting
Brief Title: Stroke-induced Immunodepression in Neurorehabilitation
Acronym: NeuroLympho
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroLympho
Record Dates: First submitted 2023-01-19; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Lymphopenia; Immunosuppression
Keywords: Ischemic stroke; Intracerebral hemorrage; Neurological rehabilitation; Neurorehabilitation; Cerebrovascular disorders; Immunodepression
MeSH Terms: conditions — Stroke; Lymphopenia; Ischemic Stroke; Cerebrovascular Disorders | interventions — Neurological Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients with immunosuppression: Patients with ischemic or hemorrhagic stroke with a neutrophil to lymphocyte ratio >= 5 at hospital admission
  Interventions: Other: Neurorehabilitation
- Stroke patients without immunosuppression: Patients with ischemic or hemorrhagic stroke with a neutrophil to lymphocyte ratio < 5 at hospital admission
  Interventions: Other: Neurorehabilitation

INTERVENTIONS:
Other: Neurorehabilitation — Four to eight weeks motor rehabilitation (500 minutes per week across 6 day per week)

SUMMARY:
The close interconnection between nervous system and the immune system is well known. Brain injuries lead to homeostasis disruption. On the one hand they result in increased brain inflammation contributing to tissue repair, at the expense of a possible extension of tissue damage. On the other hand, they lead to systemic down-regulation of innate and adaptive immunity, determining higher vulnerability to infections, responsible of death and comorbidities in the acute and subacute setting.

Aim of the study was to evaluate the role of immunosuppression in the neurorehabilitation pathway in patients with stroke.

DETAILED DESCRIPTION:
The perfect balance between nervous and immune system could be severely impaired after brain injuries, such as strokes.

In the acute phase, inflammatory mediators are responsible of central nervous system inflammation, associated to tissue repair at the expense of possible secondary brain injury or damage expansions.

In the mean time, activation of hypothalamic-pituitary-adrenal axis and the autonomic nervous system determine downregulation of innate and adaptive immunity, with decreased circulating T cell count and reduced lymphocytic response. The degree of these changes is linked to the severity of brain damage and inevitably lead to higher vulnerability to infections, representing a negative prognostic factor in the acute phase.

Association between immunosuppression and functional outcome in the neurorehabilitation setting are missing.

Aim of this study was to evaluate the role of immunosuppression in the neurorehabilitation journey in patients with stroke.

We analyzed the neutrophil-to-lymphocyte ratio, a useful tool to investigate alterations in both the innate and adaptive immune systems. We correlated it to clinical and neurorehabilitation scales, investigating disability, functional status, as well as gait analysis and occurrence of infectious complications. All outcomes were measured on admission in Neurorehabilitation setting and at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first episode of ischemic stroke or primary spontaneous intracerebral haemorrhage (both confirmed by proper neuroimaging)
* admission to the Neurorehabilitation ward within 30 days from the index event

Exclusion Criteria:

* medical history of immunodeficiency or immunoproliferative disease
* immunosuppressive or immunomodulating therapy in the year before the index event
* systemic steroids in the six months before the index event
* Glasgow Coma Scale < 8 at hospital admission
* other diagnosis of neurological diseases
* missing clinical/demographic data

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were selected from a single centre cohort admitted for stroke rehabilitation at the Neurorehabilitation Unit of the IRCCS Mondino Foundation (Pavia, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Difference between group 1 and group 2 in FIM score (Functional Independence Measure) after rehabilitation | After four to eight weeks from NRB admission
  To evaluate if stroke-induced immunosuppression is a predictor of functional independence at the end of neurorehabilitation as measured by FIM score.

SECONDARY OUTCOMES:
Difference between group 1 and group 2 in NIHSS score (National Institutes of Health Stroke Scale) after rehabilitation | After four to eight weeks from NRB admission
  To evaluate if stroke-induced immunosuppression is a predictor of neurological function at the end of neurorehabilitation as measured by NIHSS score.
Difference between group 1 and group 2 in Barthel Index after rehabilitation | After four to eight weeks from NRB admission
  To evaluate if stroke-induced immunosuppression is a predictor of performances in activities of daily living at the end of neurorehabilitation as measured by Barthel Index
Difference between group 1 and group 2 in Tinetti score after rehabilitation | After four to eight weeks from NRB admission
  To evaluate if stroke-induced immunosuppression is a predictor of motor performances at the end of neurorehabilitation as measured by Tinetti score
Difference between group 1 and group 2 in Hauser Ambulation Index score after rehabilitation | After four to eight weeks from NRB admission
  To evaluate if stroke-induced immunosuppression is a predictor of motor performances at the end of neurorehabilitation as measured by Hauser Ambulatory Index
Difference between group 1 and group 2 in infectious complication during rehabilitation | After four to eight weeks from NRB admission
  To evaluate if stroke-induced immunosuppression is a predictor of infectious complications during neurorehabilitation, namely: pneumonia (diagnosed in subjects with typical symptoms of respiratory infection, confirmed by chest X-ray abnormalities), urinary tract infections (diagnosed with a positive urine culture without evidence of contamination), sepsis (defined as acute organ dysfunction with evidence of a clear source of infection and isolation of specific pathogens on blood cultures without evidence of contamination) and other infectious complications (as gastrointestinal and skin infections)

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Science & Neurorehabilitation Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Raw data will be uploaded in the online Zenodo platform and available to other Researches upon reasonable request.

REFERENCES:
- [Result] Meisel C, Schwab JM, Prass K, Meisel A, Dirnagl U. Central nervous system injury-induced immune deficiency syndrome. Nat Rev Neurosci. 2005 Oct;6(10):775-86. doi: 10.1038/nrn1765. PMID 16163382
- [Result] Shi K, Wood K, Shi FD, Wang X, Liu Q. Stroke-induced immunosuppression and poststroke infection. Stroke Vasc Neurol. 2018 Jan 12;3(1):34-41. doi: 10.1136/svn-2017-000123. eCollection 2018 Mar. PMID 29600006
- [Result] Chamorro A, Meisel A, Planas AM, Urra X, van de Beek D, Veltkamp R. The immunology of acute stroke. Nat Rev Neurol. 2012 Jun 5;8(7):401-10. doi: 10.1038/nrneurol.2012.98. PMID 22664787
- [Result] Morotti A, Marini S, Jessel MJ, Schwab K, Kourkoulis C, Ayres AM, Gurol ME, Viswanathan A, Greenberg SM, Anderson CD, Goldstein JN, Rosand J. Lymphopenia, Infectious Complications, and Outcome in Spontaneous Intracerebral Hemorrhage. Neurocrit Care. 2017 Apr;26(2):160-166. doi: 10.1007/s12028-016-0367-2. PMID 28004330
- [Result] Wartenberg KE, Stoll A, Funk A, Meyer A, Schmidt JM, Berrouschot J. Infection after acute ischemic stroke: risk factors, biomarkers, and outcome. Stroke Res Treat. 2011;2011:830614. doi: 10.4061/2011/830614. Epub 2011 Jun 12. PMID 21789273
- [Derived] Vaghi G, Morotti A, Piella EM, Avenali M, Martinelli D, Cristina S, Allena M, Grillo V, Corrado M, Bighiani F, Cammarota F, Antoniazzi A, Ferrari F, Mazzacane F, Cavallini A, Pichiecchio A, Rognone E, Martinis L, Correale L, Castiglia SF, Trabassi D, Serrao M, Tassorelli C, De Icco R. The role of stroke-induced immunosuppression as a predictor of functional outcome in the neurorehabilitation setting. Sci Rep. 2024 Apr 9;14(1):8320. doi: 10.1038/s41598-024-58562-1. PMID 38594322